CLINICAL TRIAL: NCT05398562
Title: Simple Blind, Placebo Controlled, Randomized, Two-stage, Prospective, Single-center Safety, Tolerability and Reactogenicity Trial of the [Recombinant Tuberculosis Allergen in Standard Dilution], Solution for Intradermal Injection, 0.1 mL/Dose, Produced by FSUE SPbSRIVS FMBA of Russia, in Healthy Volunteers After a Single Dose in the Dilution of 0.1 µg / 0.1 mL or 0.2 µg / 0.1 mL
Brief Title: Tolerability and Reactogenicity Trial of the Recombinant Tuberculosis Allergen in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ATR-I-004-2019
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Tuberculosis; Skin Tests
Keywords: Tuberculosis; Diagnosis; Recombinant Tuberculosis Allergen; Mycobacterial recombinant allergens; Allergen; SPbSRIVS
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RTA / 0.1 μg / 0.1 mL (Experimental): at stage I - 5 healthy volunteers; at stage II - 20 healthy volunteers. frequency and route of administration: once, intradermally
  Interventions: Diagnostic Test: Mycobacterial recombinant allergens 0.1 μg
- RTA / 0.2 μg / 0.1 mL (Experimental): at stage I - 5 healthy volunteers; at stage II - 20 healthy volunteers. frequency and route of administration: once, intradermally
  Interventions: Diagnostic Test: Mycobacterial recombinant allergens 0.2 μg
- Placebo / 0.1 mL (Placebo Comparator): at stage I - 5 healthy volunteers; at stage II - 20 healthy volunteers. frequency and route of administration: once, intradermally
  Interventions: Diagnostic Test: Placebo

INTERVENTIONS:
Diagnostic Test: Mycobacterial recombinant allergens 0.1 μg — solution for intradermal injection, 0.1 µg / 0.1 mL
  Other Names: Recombinant tuberculosis allergen in standard dilution
  Arms: RTA / 0.1 μg / 0.1 mL
Diagnostic Test: Mycobacterial recombinant allergens 0.2 μg — solution for intradermal injection, 0.2 µg / 0.1 mL
  Other Names: Recombinant tuberculosis allergen in standard dilution
  Arms: RTA / 0.2 μg / 0.1 mL
Diagnostic Test: Placebo — solution for intradermal injection
  Arms: Placebo / 0.1 mL

SUMMARY:
Primary objective of the trial is to study the safety and tolerability of the Recombinant tuberculosis allergen in standard dilution in healthy volunteers after a single dose.

Additional trial purpose: evaluation of the product reactogenicity.

DETAILED DESCRIPTION:
The trial product is an Intradermal test to diagnose tuberculosis infection and nontuberculosis mycobacteriosis in combination with other methods. The trial will include 2 stages (stage I, II). At stage I 5 healthy volunteers will be consequently included in each group to evaluate tolerance and reactogenicity. Time required to evaluate the tolerance and reactogenicity for the first 5 volunteers in each group is less than 3 days. If no SAEs which have a "possible", "probable" and "definite" causal relationship with the product administration are observed in more than three volunteers from each group, the remaining volunteers will be allowed to take part in the trial. At stage II 20 healthy volunteers will be included in each group. Each volunteer will be assigned a two-digit randomization number.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of the volunteer's written consent to participate in the trial according to the existing legislation.
2. Age between 18 and 50 years old, inclusively.
3. Body mass index (BMI) within the range of 18.5 ≤ BMI ≤ 30 kg/m2 with body weight at least 45 kg and not more than 100 kg.
4. Verified "healthy" status: no deviations from reference values of standard clinical, laboratory and instrumental examinations. For female volunteers: negative pregnancy test (for female volunteers with preserved reproductive capacity, i.e. those who are not in menopause and who have not undergone sterilization surgery).
5. Absence of tuberculosis (TB) at chest X-ray or photofluorography
6. Negative result of TB laboratory examination (T-SPOT.TB test, sputum examination for mycobacterium tuberculosis (MBT)).
7. Negative test for HIV 1 and 2, syphilis (RPR), hepatitis В (HBsAg) and С (HCV RNA) markers.
8. Consent of the volunteer (including a female partner) to use adequate contraception methods throughout the trial and 7 days upon its completion. If hormonal contraceptives are used, they must be canceled at least 2 months before the start of the trial.
9. Hemodynamic and other vital signs should be within normal limits (reference intervals are 60-90 beats/min at rest for heart rate (HR), up to 22 per minute for respiratory rate (RR), body temperature (BT) from 35.5 to 36.9 °C; systolic blood pressure (SBP) is considered normal blood pressure (BP) in the range of 100-130 mmHg, diastolic blood pressure (DBP) is considered normal in the range of 60-89 mmHg).
10. Negative breath alcohol test.
11. Negative urinalysis for abuse of medicinal products (MP) and consumption of narcotic substances (NS), including cocaine, cannabis, amphetamies, barbiturates and opiods.
12. Abstinence from alcohol for 14 days before the start of the trial and until the end of participation in the trial.
13. Abstinence from smoking for 48 hours before the start of the trial and during hospitalization.

Exclusion Criteria:

1. Inability to provide an informed consent.
2. History of allergies.
3. Acute or chronic infectious diseases (including flu, ARVI) within 30 days before the start of the trial.
4. History of tuberculosis or known contact of a volunteer and/or their family members with a person infected with TB.
5. Contact with MBT carriers.
6. Symptoms of pulmonary or extrapulmonary TB, respiratory and systemic TB.
7. Symptoms of mycobacteriosis (chronic productive cough, asthenia, fever, sweating) and/or changes (infiltration with degradation, nodules, tumor like lesions) at chest X-ray/photofluorography during screening or according to the medical history.
8. Congenital or acquired abnormalities of the immune system.
9. A history of diseases affecting lymphoid organs (Hodgkin lymphoma, other lymphomas, leukemias, sarcoidosis).
10. A history of epilepsy.
11. Viral or bacterial infection that may affect cellular immune response during the screening.
12. Generalized skin diseases, including eczema, psoriasis, ichthyosis, burns, rash etc.
13. A condition affecting the blood clotting and causing a risk of hemorrhage.
14. Any immunomodulatory therapy (immunoglobulins, systemic corticosteroids, methotrexate, azathioprine, cyclosporine, infliximab and other blood products) 6 months before the start of the trial.
15. Previous vaccination 6 months before the start of the trial.
16. Consumption of medicinal products that have a significant impact on hemodynamics, liver function etc. (barbiturates, omeprazole, cimetidine etc.), oral anticoagulants, products metabolized by CYP2D6 less than 2 months before the start of the trial.
17. Vital signs outside the reference ranges: SBP less than 100 mmHg or more than 130 mmHg; DBP less than 60 mmHg or more than 89 mmHg; HR less than 60 bpm or more than 90 bpm; BT less than 35.5 or more than 36.9°С, RR more than 22 breaths per minute.
18. Laboratory values outside the reference ranges.
19. TB foci at chest X-ray or photofluorography.
20. Positive result of TB laboratory examination (T-SPOT.TB test, sputum examination for MBT).
21. Tuberculin skin test (Mantoux test) or Diaskintest less than 6 months before the start of the trial.
22. Consumption more than 5 units of alcohol per week (where each unit is equal to 30 mL of strong drinks or 325 mL of beer) and/or a history of alcohol, product, substance abuse and abuse of medicinal products.
23. Smoking more than 10 cigarettes per day and inability to refrain from smoking 48 hours before the start of the trial and during the hospital stay.
24. Special diet (e.g. vegetarian, vegan, with limited salt consumption) or life style (night shifts, extreme physical efforts).
25. Positive breath alcohol test.
26. Positive urinalysis for MP abuse and consumption of narcotic substances (NS), including cocaine, cannabis, amphetamies, barbiturates and opiods.
27. Positive pregnancy test, lactation period (for female volunteers).
28. Donation (450 or more mL of blood) within 30 days before the start of the trial.
29. Participation in any phase of the clinical trial 90 days before the start of the trial.
30. Unavailability for observation throughout the trial, inability to comply with the visit schedule, inability to be hospitalized for a period of up to 5.5 days, high risk of problems that may occur during the central line installation or upper arm vein puncture.
31. Affiliation with the vulnerable group of volunteers (minors; incapable persons; people with limited freedom of expression or people who might be participating in the trial against their will (serving sentences, held in detention, military personnel).
32. Other reasons which, in the investigator's opinion, prevent the volunteer to take part in the trial or create an unjustified risk.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | Days 0 - 15

SECONDARY OUTCOMES:
Number of participants with abnormal changes in laboratory parameters - Complete blood count (CBC) | Days 0, 1; 72 hours upon the administration, day 15
  hemoglobin, red blood cells, hematocrit, thrombocytes, leukocytes, ESR, differential leukocyte count (neutrophils, lymphocytes, eosinophils, monocytes, basophils)
Number of participants with abnormal changes in laboratory parameters - Biochemical blood test (BBT) | Days 0, 1; 72 hours upon the administration, day 15
  total protein, creatinine, urea, glucose, total bilirubin, direct bilirubin, ALT, AST, AP, CRP, total LDH, total cholesterol, PTI
Number of participants with abnormal changes in laboratory parameters - Immunologic blood test (IBT) | Days 0, 1; 72 hours upon the administration, day 15
  IgA,IgM, IgG and IgE in blood serum
Number of participants with abnormal Changes in laboratory parameters - Urinalysis (UA) | Days 0, 1; 72 hours upon the administration, day 15
  color, transparency, pH, specific gravity, nitrites, protein, glucose, ketones, urobilinogen, bilirubin, microscopic examination: erythrocytes, leukocytes, casts, except for hyaline casts, bacteria
Number of participants with abnormal ECG findings | Days 0, 1; 72 hours upon the administration, day 15
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1 - V6)
Number of participants with abnormal changes in physical examination data | Days 0, 1; 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 hours after administration, day 15
  Physical examination includes examination of skin and visible mucous membranes, assessment of musculoskeletal system, lymph node palpation, thyroid palpation, objective examination of organ systems (cardiovascular, respiratory, digestive, urinary systems, ear, nose, throat, auscultation of heart and lungs, abdominal examination (sizes of liver and spleen), examination of kidneys, central nervous system)
Number of participants with abnormal changes in the functions of vital organs and vital signs - Heart rate (HR) | Days 0, 1; 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 hours after administration, day 15
  The HR is measured during auscultation of the heart in parallel with determining the pulse rate on the radial artery (or on the carotid artery in case of weak pulsation in the radial artery) for a minute while sitting/lying.
Number of participants with abnormal changes in the functions of vital organs and vital signs - Respiratory rate (RR) | Days 0, 1; 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 hours after administration, day 15
  RR is measured for a minute at rest in the seated/supine position, by registering the breathing movements of the chest or abdominal wall, without attracting the volunteer's attention.
Number of participants with abnormal changes in the functions of vital organs and vital signs - Blood pressure (BP): Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) | Days 0, 1; 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 hours after administration, day 15
  BP (SBP and DBP) is measured on the brachial artery in the prone position according to the Korotkoff method using a certified instrument to measure BP on the same arm with a cuff of length and width matching the length and circumference of the volunteer's shoulder in accordance with the BP measurement recommendations.
Number of participants with abnormal changes in the functions of vital organs and vital signs - Body temperature (BT) | Days 0, 1; 20 min. (00:20), 2, 5, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 hours after administration, day 15
  BT is measured with a mercury or digital thermometer in the armpit for at least 5 minutes.
Incidence and severity of immediate hypersensibility reactions in each group according to the four-point scale | 20 minutes, 2, 5, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 hours after the administration, day 15
  * Pruritus at the site of TP/RP injection;
  * Burning sensation at the site of TP/RP injection.
  The assessment will be carried out according to the four-point scale:
  * 0 - no symptoms;
  * 1 - mild symptoms;
  * 2 - symptoms that significantly disrupt normal daily activities;
  * 3 - symptoms that cancel normal daily activities.
Proportion of volunteers who have withdrawn from the trial early due to the AE/SAE | Days 0 - 15
Incidence of systemic post-injection reactions | 20 minutes, 2, 5, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 hours after the administration, day 15
  * Fever;
  * Cough;
  * Pharyngitis;
  * Fatigue;
  * Arthralgias;
  * Myalgias;
  * Headache;
  * Diarrhea;
  * Chills.
  the four-point scale:
  * 0 - no symptoms;
  * 1 - mild symptoms;
  * 2 - symptoms that significantly disrupt normal daily activities;
  * 3 - symptoms that cancel normal daily activities.
Incidence of local post-injection reactions | 20 minutes, 2, 5, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 hours after the administration, day 15
  * Hyperemia at the injection site;
  * Soreness;
  * Tumidity;
  * Swelling/infiltrate;
  * Enlarged regional lymph nodes;
  * Mucosal changes, papula, vesicle, erosion.
  the four-point scale:
  * 0 - no symptoms;
  * 1 - mild symptoms;
  * 2 - symptoms that significantly disrupt normal daily activities;
  * 3 - symptoms that cancel normal daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Limited Liability Company "Scientific Research Center Eco-Safety", Saint Petersburg, Russia